CLINICAL TRIAL: NCT03354533
Title: Study of ORL-1F (L-fucose) in Patients With Leukocyte Adhesion Deficiency Type II
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orpha Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ladtwo-1
Record Dates: First submitted 2017-11-21; First posted 2017-11-28 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Leukocyte Adhesion Deficiency, Type II
MeSH Terms: conditions — Congenital disorder of glycosylation, type 2C | interventions — Fucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | US Export: No

ARMS (1):
- Treatment with ORL-1F - L-fucose (Other)
  Interventions: Drug: L-fucose

INTERVENTIONS:
Drug: L-fucose — Oral ORL-1F

SUMMARY:
Study of ORL-1F in Patients With Leukocyte Adhesion Deficiency Type II

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Leukocyte Adhesion Deficiency Type II.
* Less than 18 years old.

Exclusion Criteria:

* Diagnosis of any other disease that is not a manifestation of Leukocyte Adhesion Deficiency Type II.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Decrease in infection frequency | 12 months after treatment started
  Statistically significant decrease in infection frequency

SECONDARY OUTCOMES:
Decrease in neutrophil count | 30 days after treatment started
  Statistically significant decrease in absolute neutrophil count

IPD SHARING:
Plan to Share IPD: No